CLINICAL TRIAL: NCT02670772
Title: A Randomised, Double-Blind, Multi-Centre, Parallel-Group Phase 3b Study to Demonstrate Non-inferiority of Stavudine (20 mg Twice Daily) Compared With Tenofovir Disoproxil Fumarate (300 mg Once Daily) When Administered in Combination With Lamivudine and Efavirenz in Antiretroviral-Naive Patients Infected With HIV-1
Brief Title: Dose Optimisation of Stavudine for the Treatment of HIV Infection
Acronym: D4T
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Willem Daniel Francois Venter (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor-Investigator, Willem Daniel Francois Venter, Professor, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WRHI001; BMGF (Other Grant/Funding Number: OPP1032239)
Record Dates: First submitted 2016-01-22; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Acquired Immune Deficiency Syndrome; Human Immunodeficiency Virus
Keywords: Antiretroviral Agents
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Stavudine; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stavudine (Active Comparator): Stavudine 20mg twice daily for 96 weeks
  Interventions: Drug: Stavudine
- Tenofovir Disoproxil Fumarate (Active Comparator): Tenofovir 300mg once daily for 96 weeks
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Stavudine — Stavudine 20mg twice daily for 96 weeks + Placebo 300mg once daily for 96 weeks + Lamivudine 150mg twice daily for 96 weeks + Efavirenz 600mg once daily for 96 weeks
  Other Names: d4t
  Arms: Stavudine
Drug: Tenofovir Disoproxil Fumarate — TDF 300mg once daily + Placebo 20mg twice daily for 96 weeks + Lamivudine 150mg twice daily for 96 weeks + Efavirenz 600mg once daily for 96 weeks
  Other Names: TDF
  Arms: Tenofovir Disoproxil Fumarate

SUMMARY:
The purpose of this study is to demonstrate whether low dose stavudine (d4T) is non-inferior (in terms of both viral suppression and toxicity) to tenofovir (TDF) after 2 years of HIV treatment.

DETAILED DESCRIPTION:
This is randomised, placebo-controlled, double-blind, parallel-group, multisite, study to demonstrate whether low dose stavudine (d4T) is non-inferior to tenofovir (in terms of both viral suppression and toxicity) to tenofovir (TDF) after 2 years of HIV treatment. If so, this will allow approximately two people requiring antiretrovirals to be treated for the price of one, with the same outcomes at two years. This is of huge public health consequence in Southern Africa, where TDF and zidovudine (AZT) now consume the majority of the antiretroviral budget. Decreasing total drug doses of antiretroviral agents, while maintaining efficacy, represents an untapped possibility for decreasing costs and toxicity, if efficacy can be maintained. Stavudine (d4T), an NRTI, is currently the second most commonly used antiretroviral worldwide in developing countries. Stavudine is an ideal candidate for assessment because of low cost, widespread use, and co-formulation, albeit at a dose that has significant side effects. While well tolerated in the short term, dose-dependent medium and long-term side effects, namely lipoatrophy and peripheral neuropathy, are very common. lipoatrophy is insidious, largely irreversible, and highly stigmatising, These toxicities have lead to the withdrawal of Stavudine as a recommended drug in most countries that can afford an alternative, even in second and subsequent regimens; the World Health Organisation (WHO) recommends that countries, wherever possible, move away from using Stavudine. However, there are data that suggest a lower dose of Stavudine would be better tolerated than the currently recommended dose and will be as effective in suppressing viral load as currently preferred first-line drugs. Consented patients will be randomised into one of two treatment arms using the interactive voice response systems (IVRS). The study monitor will maintain current personal knowledge of the study through observation, review of study records and source documentation, and discussion of the conduct of the study with the principal investigator or sub investigator and staff. Data will be captured onto electronic data capture system and managed for completeness, consistency and accuracy. All study operations such as patient recruitment, data management, safety reporting will be guided by Standard Operating Procedure (SOP) documents. A total of 1068 male and female antiretroviral-naive patients infected with HIV-1 will be randomised in a 1:1 ratio (approximately 534 patients per treatment group) to Treatment Group 1 (d4T/3TC+EFV) or Treatment Group 2 (TDF/3TC+EFV). Approximately 15% of patients are expected not to be evaluable for the PP set, therefore resulting in 907 patients for the PP set. This will provide 90% power to show non-inferiority between the 2 treatment groups for the proportion of patients achieving the primary efficacy endpoint (undetectable plasma HIV-1 RNA levels [<50 copies/mL] at Week 48) for the PP set (and 94% power for the all-randomised set), using a non-inferiority margin of 10% and a 1-sided 2.5 significance level. The proportion of patients achieving the primary efficacy endpoint has been assumed to be 70% in both treatment groups. The sample size calculation has been adjusted to allow for stopping at 2 interim analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female aged ≥18 years (upper limit of <65 years in India)
* Patient has a documented laboratory diagnosis of infection with HIV-1 (positive enzyme-linked immunosorbent assay HIV-1 antibody test) at screening or from previous records
* Patient has a life expectancy of ≥2 years in the opinion of the investigator
* Patient has a plasma HIV-1 RNA level >1000 copies/mL
* Patient has a plasma CD4 count ≤ 350 cells/mm3 using standard flow cytometry.
* Patient has the following clinical chemistry and haematological laboratory results:

  * Serum creatinine ≤1.5 mg/dL (133 μmol/L) and a calculated creatinine clearance level ≥60 mL/min according to the Cockcroft-Gault formula
  * Serum alanine aminotransferase <5 × upper limit of normal (ULN)
  * Serum aspartate aminotransferase <5 × ULN
  * Serum lipase ≤1.5 × ULN
  * Total bilirubin ≤1.5 mg/dL (25 μmol/L) unless felt by clinician to be due to Gilbert syndrome
  * Haemoglobin ≥7.0 g/dLAbsolute neutrophil count ≥500/mm3
  * Platelet count ≥50 000/mm3.
* Female patients of childbearing potential, including those who are less than 2 years post-menopausal, must agree to, and comply with using a highly effective method of birth control (eg, barrier contraceptives [condom or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectable, combination oral contraceptives, transdermal patches, or contraceptive rings], intrauterine devices, or sexual abstinence) while participating in this study. In addition, all women of childbearing potential must agree to continue to use birth control throughout the study until last study visit Women Not of Childbearing Potential are women who are postmenopausal or permanently sterilised (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy).
* Women of Childbearing Potential (WOCBP) - Any female who has experienced menarche and does not meet the criteria for "Women Not of Childbearing Potential".
* Patient has the ability to comprehend the full nature and purpose of the study, in the opinion of the investigator, including possible risks and side effects, to cooperate with the investigator, to understand verbal and written instructions, and to comply with the requirements of the entire study
* Patient is informed of the full nature and purpose of the study, including possible risks and side effects, given ample time and opportunity to read and understand this information, and sign and date the written informed consent before inclusion in the study

Exclusion Criteria:

* Patients who have previously received treatment with any form of antiretroviral therapy, including preventing mother-to-child transmission regimens
* Patients who are taking and cannot discontinue the following prohibited concomitant medications at least 1 week prior to the baseline visit and for the duration of the study period:

  * Any agents with significant nephrotoxic potential
  * Probenecid
  * Systemic chemotherapy agents
  * Drugs that have significant interactions with EFV other than rifampicin Administration of any of the above medications should be discontinued at least 1 week prior to the baseline visit and for the duration of the study period.
* Patients who are clinically unstable, in the investigator's opinion, should be stabilized prior to inclusion into this study and their baseline concomitant medications should be stable for at least 1 month (30 days) prior to enrolment. In addition, investigators should not anticipate changing dose levels or medications for the duration of the study. Patients who, in the investigator's opinion, require HIV-related prophylaxis (such as cotrimoxazole) and/or other HIV-related treatments (e.g. treatment for oral thrush, tuberculosis, etc) and who, in the investigator's opinion are clinically stable may have such treatment initiated or discontinued during the screening period. The 30-day waiting period will not apply to the latter.
* Patients who have a current history of drug or alcohol abuse that, in the opinion of the investigator, may be an impediment to patient adherence to the protocol
* Patients who have a medical history or evidence of gastrointestinal malabsorption syndrome, chronic nausea, or vomiting which may prevent patients receiving oral medication
* Patients who have participated in a study with an investigational drug within 60 days of screening or who are currently receiving treatment with any other investigational drug or device
* Patients who are hepatitis B surface antigen positive
* Patients with symptomatic peripheral neuropathies
* Female patients who are currently pregnant or breastfeeding
* Female patients desiring pregnancy during the next 2 years
* Patients who have a strong likelihood of relocating far enough to make access to the study site difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1077 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with undetectable plasma HIV-1 RNA levels | Week 48
Number of participants with adverse events related to treatment | Week 48

SECONDARY OUTCOMES:
Number of patients with plasma HIV-1 RNA levels <200 copies | Week 96
Number of participants with abnormal Bone mineral density and fat distribution | Week 96
Number of participants with abnormal Bone mineral density. | Week 96
Number of participants with abnormal fat distribution | Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Francois Venter, FCP (SA), Principal Investigator — Wits Reproductive Health & HIV Institute
Locations (3):
- VHS-YRG Care Medical Centre, Chennai, Tamil Nadu, India
- Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng, South Africa
- The Infectious Disease Institute (IDI), Mulago Hospital Complex, Kampala, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Draaijer M, Lalla-Edward ST, Venter WDF, Vos A. Phone Calls to Retain Research Participants and Determinants of Reachability in an African Setting: Observational Study. JMIR Form Res. 2020 Sep 30;4(9):e19138. doi: 10.2196/19138. PMID 32996891
- [Derived] Venter WDF, Kambugu A, Chersich MF, Becker S, Hill A, Arulappan N, Moorhouse M, Majam M, Akpomiemie G, Sokhela S, Poongulali S, Feldman C, Duncombe C, Ripin DHB, Vos A, Kumarasamy N. Efficacy and Safety of Tenofovir Disoproxil Fumarate Versus Low-Dose Stavudine Over 96 Weeks: A Multicountry Randomized, Noninferiority Trial. J Acquir Immune Defic Syndr. 2019 Feb 1;80(2):224-233. doi: 10.1097/QAI.0000000000001908. PMID 30640204
- [Derived] Vos AG, Chersich MF, Klipstein-Grobusch K, Zuithoff P, Moorhouse MA, Lalla-Edward ST, Kambugu A, Kumarasamy N, Grobbee DE, Barth RE, Venter WD. Lipid levels, insulin resistance and cardiovascular risk over 96 weeks of antiretroviral therapy: a randomised controlled trial comparing low-dose stavudine and tenofovir. Retrovirology. 2018 Dec 14;15(1):77. doi: 10.1186/s12977-018-0460-z. PMID 30547820